CLINICAL TRIAL: NCT06988683
Title: Investigation of Posture, Core Stabilization, Respiratory Muscle Strength and Function, and Quality of Life in Women With Urinary Incontinence
Brief Title: Posture, Core Stabilization, Respiratory Muscle Strength and Quality of Life in Women With Urinary Incontinence
Status: Completed | Type: Observational
Sponsor: Izmir Democracy University (Other)
Responsible Party: Principal Investigator, Özlem Çınar Özdemir, Prof.Dr, Izmir Democracy University
Other Study IDs: urinary incontinence
Record Dates: First submitted 2025-01-15; First posted 2025-05-25 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Urinary Incontinence (UI)
Keywords: Core stabilization; cough force; posture; respiratory muscle strength; urinary incontinence; maximal expiratory pressure
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study Group (Urinary incontinance): The study included 32 volunteer individuals who were diagnosed with urinary Incontinance and fulfilled the inclusion criteria.
  Pad test was applied to evaluate the degree of urinary incontinence of the patients. Posture analyses of the individuals were evaluated with Fizyosoft Becure Mobile Posture Application. Stabiliser Pressure Biofeedback Unit® (BBU) (Chattanooga Medical Suplly Inc, Chattanooga, TN) was used for core muscle stabilisation, Cosmed® Pony FX was used for respiratory muscle strength and functions and ExpiRite Peak Flow Meter (ExpiRite Peak Flow Meter, China) was used for cough strength assessment. Modified Constipation Rating Scale (MCAS), Rome IV Criteria, Bristol Stool Scale (BGS) were used to evaluate constipation, while quality of life and pelvic floor symptoms were evaluated using Urogenital Distress Inventory (UDI-6), Incontinence Impact Questionnaire (IIQ-7) and Global Pelvic Floor Discomfort Questionnaire (GPTRA).
- Control Group: The study included 30 asymptomatic volunteers without urinary incontinence without a diagnosis of UI.
  In this study, demographic information form was used to evaluate the socio-demographic status. Posture analyses of the individuals were evaluated with Fizyosoft Becure Mobile Posture Application. Stabiliser Pressure Biofeedback Unit® (BBU) (Chattanooga Medical Suplly Inc, Chattanooga, TN) was used for core muscle stabilisation, Cosmed® Pony FX was used for respiratory muscle strength and functions and ExpiRite Peak Flow Meter (ExpiRite Peak Flow Meter, China) was used for cough strength assessment. Modified Constipation Rating Scale (MCAS), Rome IV Criteria, Bristol Stool Scale (BGS) were used to evaluate constipation, while quality of life and pelvic floor symptoms were evaluated using Urogenital Distress Inventory (UDI-6), Incontinence Impact Questionnaire (IIQ-7) and Global Pelvic Floor Discomfort Questionnaire (GPTRA).

SUMMARY:
When the literature was examined, it was observed that there were studies on parameters such as quality of life, pelvic floor muscle strength in women with urinary incontinence, but there were not enough studies on posture, respiratory function, constipation and cough strength. Therefore, in this study, the researchers aimed to investigate posture, constipation, core muscle stabilisation, respiratory muscle strength and function, cough strength and quality of life of women with urinary incontinence and to compare these parameters with women without urinary incontinence.

DETAILED DESCRIPTION:
Urinary incontinence (UI) is involuntary urinary leakage and may lead to social and economic problems. There are different types of UI such as stress type, urge, mixed type. Risk factors include age, gender, genetics, menopause, obesity, labour and surgical history. Posture is the position of the body during movement or posture and can also be defined as muscle balance. Studies have reported that there may be a relationship between UI and respiratory problems and postural motor control disorder. Various methods are used in posture assessment, but there is no study evaluating posture with artificial intelligence in women with UI in the literature.Constipation is a particularly serious risk for the development of stress urinary incontinence (SUI). Severe constipation in women leads to differences in the neural function of the pelvic floor by reducing the neural effect of the external anal sphincter and pelvic floor muscles (PFM). Many conditions that increase intra-abdominal pressure (IAB) cause the onset or development of UI. Constipation also leads to an increase in intra-abdominal pressure and thus an increase in intra-bladder pressure. Recently, researchers have investigated the relationship between constipation and urinary incontinence, but the results have been inconsistent. Core stabilisation is the ability to regulate the posture and movement of the body over the pelvis. During forced exhalation activities (Valsalva, coughing, laughing, etc.), the pelvic floor muscles (PFM), abdominal muscles and diaphragm work together to increase intra-abdominal pressure and prevent incontinence. The trunk stabilisation muscles work in concert to keep the abdomen and lumbopelvic region stable by regulating intra-abdominal pressure during various activities of daily living. The activity of these muscles alters intra-abdominal pressure, which in turn can affect the activity of the pelvic floor muscles. Cough is associated with urinary incontinence in women by affecting the concerted contraction of thoracic, abdominal and pelvic muscles. Women with chronic cough are 55-63.3% more likely to develop severe UI than women without chronic cough. Chronic cough has been shown to be one of the common risk factors for UI, along with advanced age, high BMI, history of vaginal delivery and surgical interventions. Urinary incontinence is a public health problem that seriously affects women's quality of life and social participation, as well as being common among older women. UI has a negative impact on individuals' sleep, sexual function, work performance and psychosocial aspects. As symptoms increase, quality of life decreases, but women usually realise the effects of UI years later by seeking professional help. When the literature was reviewed, it was observed that there were studies on parameters such as quality of life and pelvic floor muscle strength in women with urinary incontinence, but there were not enough studies on posture, respiratory functions, constipation and coughing strength. Therefore, in this study, the researchers aimed to investigate posture, constipation, core muscle stabilisation, respiratory muscle strength and function, cough strength and quality of life of women with urinary incontinence and to compare these parameters with women without urinary incontinence.

ELIGIBILITY:
Inclusion Criteria:

1. Inclusion Criteria for Women with Urinary Incontinence

   * Being diagnosed with urinary incontinence
   * Volunteer to participate in the study
   * To be over 18 years of age
   * To be able to communicate verbally and in written Turkish
2. Inclusion Criteria for Women without Urinary Incontinence

   * No symptoms of urinary incontinence
   * Volunteer to participate in the study
   * To be over 18 years of age
   * Establish written and verbal communication in Turkish

Exclusion Criteria:

* The presence of any pathology that may affect pelvic floor function
* Trauma to the lumbopelvic, abdominal, thoracic or lower extremities within the last six months
* Urinary tract infection
* Grade III or higher urogenital prolapse
* Neurological or psychiatric illness
* Being pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: This study, in which we aimed to evaluate individuals diagnosed with urinary incontinence, was conducted in the Gynaecology and Obstetrics outpatient clinic of Buca Seyfi Demirsoy Training and Research Hospital. Individuals diagnosed with UI by an Obstetrics and Gynaecology Specialist were included in the study. Thirty-two volunteer individuals diagnosed with UI who met the inclusion criteria and 30 individuals without urinary incontinence were included in the study.
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-06-24 (Actual)

PRIMARY OUTCOMES:
Maximal inspiratory pressure (MIP) | 1 year
  The MIP which shows respiratory muscle strength will be evaluated using a portable mouth pressure measuring device based on American Thoracic Society and European Respiratory Society criteria.
Maximal expiratory pressure (MEP) | 1 year
  The MEP which shows respiratory muscle strength will be evaluated using a portabl mouth pressure measuring device based on American Thoracic Society and European Respiratory Society criteria.

SECONDARY OUTCOMES:
Forced vital capacity (FVC) | 1 year
  Pulmonary function (Forced vital capacity (FVC)) will be evaluated with a spirometer. In the study, measurements will be made using the Cosmed Omnia microQuark 1.5 (Cosmed, Rome, Italy) device. Considering that dizziness may occur during forced expiration, measurements will be made while individuals are in a sitting position. While participants are sitting in a comfortable position in a chair with a backrest, nose clip will be attached and they will be asked to bite the mouthpieces with their teeth and close their lips in a way that does not allow air to escape. The tests will be performed at least 3 times by the participants and care will be taken to ensure that the expiration time is at least 6 seconds and the plateau time is 1 second. Due to the device software that records all three data, it saves the average of the two best data and processes it as a value.
Forced expiratory volume in the first second (FEV1) | 1 year
  Pulmonary function (Forced expiratory volume in the rst second (FEV1)) will be evaluated with a spirometer.
FEV1/FVC | 1 year
  Pulmonary function (FEV1/FVC) will be evaluated with a spirometer.
Flow rate 25-75% of forced expiratory volume (FEF 25-75%) | 1 year
  Pulmonary function (Flow rate 25-75% of forced expiratory volume (FEF 25-75%)) will be evaluated with a spirometer.
Peak flow rate (PEF) | 1 year
  Pulmonary function (Peak ow rate (PEF)) will be evaluated with a spirometer.
Posture Assessment | 1 year
  Posture assessment will be performed using an artificial intelligence based posture analysis package developed by Fizyosoft and Becure.
Core Stabilization Assessment | 1 year
  Stabilizer Pressure Biofeedback Unit (Chattanooga, USA) will be used for core stabilization assessment. The five-level core stabilization test developed by Sahrmann will be used to assess the participants' core stabilization levels.
Cough Force Assessment | 1 year
  Cough force will be measured using a portable peak flow meter (PEF meter) (ExpiRite Peak Flow Meter, China). During the test, participants cough vigorously into the device following a deep inspiration in an upright position. The peak flow rate (PEF) reached is recorded and a disposable mouthpiece is used for each participant. Three measurements are taken and the highest value is taken for analysis, with a 30 second rest period between measurements.
Modified Constipation Assessment Scale | 1 year
  This scale was developed by McMillan et al. in 1989 to determine the status and severity of constipation. It is a valid and reliable questionnaire consisting of nine questions and can be used in children and adults. Respondents rate each question as "no problem" (0), "some problem" (1) or "severe problem" (2). The total score ranges from zero (no constipation) to 18 (most severe constipation).
Rome IV Criteria | 1 year
  It is a clinical guideline defining the presence of constipation. The Rome IV criteria have been modified with regard to the frequency of abdominal pain, emphasizing the need for more frequent episodes of abdominal pain for diagnosis. At least two of these symptoms must occur at least once a week for a month, without any other underlying medical condition.
Bristol Stool Scale | 1 year
  Developed in 1990 by Lewis and Heaton at the University of Bristol, the Bristol Stool Scale (BGS) is a scale that assesses the physical properties and intestinal transit time of stool. Stool is divided into seven types: Types 3, 4 and 5 indicate normal stools; Types 1 and 2 indicate constipation; and Types 6 and 7 indicate diarrhea. Low scores indicate slow and high scores indicate fast intestinal transit.
Urogenital Distress Inventory (UDI-6) and Incontinence Impact Questionnaire (IIQ-7) | 1 year
  UDI-6 and IIQ-7 are short forms that assess the quality of life in urinary incontinence. The UIQ-6 consists of 6 questions including symptoms of urge, stress and emptying and the score is between 0-18. The IIQ-7 consists of 7 questions assessing physical activity, travel, social relationships and emotional health, with a score between 0-21. Higher scores indicate a reduced quality of life.
Global Pelvic Floor Bother Questionnaire | 1 year
  This questionnaire is a scale that assesses women's pelvic floor symptoms and severity. It covers symptoms such as urinary incontinence, pelvic organ prolapse and fecal incontinence. It consists of nine questions; respondents answer "yes/no" and rate severity from 1-5. The total score is 0-100, with a higher score indicating more symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Özlem Çinar Özdemir, Prof.Dr, Principal Investigator — İzmir Democracy University
Locations (1):
- Izmir Democracy University, Izmir, Karabağlar/İzmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Talasz H, Kofler M, Kalchschmid E, Pretterklieber M, Lechleitner M. Breathing with the pelvic floor? Correlation of pelvic floor muscle function and expiratory flows in healthy young nulliparous women. Int Urogynecol J. 2010 Apr;21(4):475-81. doi: 10.1007/s00192-009-1060-1. Epub 2009 Dec 8. PMID 19997721
- [Result] Stein TA, DeLancey JO. Structure of the perineal membrane in females: gross and microscopic anatomy. Obstet Gynecol. 2008 Mar;111(3):686-93. doi: 10.1097/AOG.0b013e318163a9a5. PMID 18310372
- [Result] Steenstrup B, Pelleray M, Cornu JN, Verdun S, Gilliaux M. Neutral posture education during cough can reduce urine leakage in women with cough-related stress urinary incontinence. Prog Urol. 2023 Dec;33(17):1083-1091. doi: 10.1016/j.purol.2023.09.002. Epub 2023 Sep 26. PMID 37758607
- [Result] Shi ZH, Jonkman A, de Vries H, Jansen D, Ottenheijm C, Girbes A, Spoelstra-de Man A, Zhou JX, Brochard L, Heunks L. Expiratory muscle dysfunction in critically ill patients: towards improved understanding. Intensive Care Med. 2019 Aug;45(8):1061-1071. doi: 10.1007/s00134-019-05664-4. Epub 2019 Jun 24. PMID 31236639
- [Result] Ptaszkowski K, Paprocka-Borowicz M, Slupska L, Bartnicki J, Dymarek R, Rosinczuk J, Heimrath J, Dembowski J, Zdrojowy R. Assessment of bioelectrical activity of synergistic muscles during pelvic floor muscles activation in postmenopausal women with and without stress urinary incontinence: a preliminary observational study. Clin Interv Aging. 2015 Sep 23;10:1521-8. doi: 10.2147/CIA.S89852. eCollection 2015. PMID 26445533